CLINICAL TRIAL: NCT05411744
Title: One-month Latent Tuberculosis Treatment for Renal Transplant Candidates
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Pinki Bhatt, Associate Professor, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro2018001735
Record Dates: First submitted 2022-06-06; First posted 2022-06-09 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Latent Tuberculosis; End Stage Renal Disease; Renal Transplant Candidate for Right Kidney; Renal Transplant Candidate for Left Kidney
Keywords: Latent Tuberculosis; End Stage Renal Disease; Renal Transplant Candidate
MeSH Terms: conditions — Latent Tuberculosis; Kidney Failure, Chronic | interventions — rifapentine; Isoniazid; Vitamin B 6

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- 1 month Rifapentine, Isoniazid and Vitamin B6 (Other): Participants will receive 28 days of self-administered daily doses of RPT, INH, and pyridoxine (vitamin B6).
  There are no multiple arms or multiple interventions. All participants will receive all 3 drugs. There are no comparators.
  Interventions: Drug: 1 month Rifapentine, Isoniazid and Vitamin B6

INTERVENTIONS:
Drug: 1 month Rifapentine, Isoniazid and Vitamin B6 — Participants will be treated with one month (4 weeks) of daily Isoniazid, Rifapentine and Vitamin B6.

SUMMARY:
This is a prospective, single-center, single-arm, open-label study investigating the safety, compliance and pharmacokinetics of 1-month treatment of Isoniazid, Rifapentine and Vitamin B6 in renal transplant candidates.

DETAILED DESCRIPTION:
Latent tuberculosis infection (LTBI) or inactive tuberculosis, is a common disease found in patients with end-stage renal disease (ESRD) who are being considered for renal transplant (RT). Approximately 5-15% of patients with LTBI will convert to an active form of TB, especially in patients with a weak immune system. Given the morbidity and mortality associated with active TB disease along with the public health threat, LTBI is routinely treated in pre-transplant candidates. While treatment with isoniazid (INH) for 9 months is the mainstay of therapy, its use poses some clinical challenges due to the prolonged duration of treatment, risk of adverse drug effects, and suboptimal compliance and treatment completion. In addition to these challenges, the consequences of delays in transplant due to the time it takes to complete current treatment options are notable. Most recently, there is a large international, randomized, prospective, phase 3 clinical trial by Swindell et al., that found that 1 month of INH and Rifapentine (1m-INH-RPT) compared to the standard 9-month regimen of INH in HIV patients with LTBI had similar TB incidence in both treatment arms but higher compliance rate and fewer adverse events for patients taking 1m-INH-RPT. Given these findings, if a similar study can be conducted in renal transplant candidate population, it can alleviate the aforementioned challenges being faced in RT candidates. Thus, this is a single-arm, open-label, prospective clinical trial investigating the safety, compliance, pharmacokinetics of 1m-INH-RPT in RT candidates.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women Age > 18
* Weight > 30 kg
* End-stage renal disease
* Living-related or deceased kidney transplant candidate (not on the waitlist) deemed by their transplant nephrologist
* Negative serum OR urine pregnancy test
* Evidence of latent tuberculosis or high risk for tuberculosis: (1) Confirmed positive tuberculin skin test (TST) ≥ 5 mm or positive quantiferon gold test/T-spot and a chest radiograph or chest CT scan without evidence of active pulmonary TB OR (2) Patients with negative TST or quantiferon gold/T-spot test but high risk for tuberculosis are eligible if they have (i) radiographic evidence of previous TB (stable fibronodular changes, including scarring [peribronchial fibrosis, bronchiectasis, and architectural distortion] and nodular opacities in the apical and upper lung zones) and no history of adequate treatment, or (ii) have had close and prolonged contact with a case of active TB.

Exclusion Criteria:

* Age <18 years
* Absolute neutrophil count of <750 cells/mm3
* Hemoglobin < 7.4 g/dL
* Platelets < 50 x 10E3/uL
* AST (SGOT) and ALT (SGPT) > 3 times the upper limit of normal (ULN)
* Total bilirubin > 2.5 times the ULN
* Presence of active TB
* Prior history of treatment for active TB or LTBI
* Known exposure to multidrug-resistant TB
* Known history of or active porphyria
* History of liver cirrhosis
* Evidence of active acute hepatitis
* Peripheral neuropathy > grade 2
* Active drug or alcohol dependence in opinion of investigator that will interfere with adherence
* On non-modifiable medications with significant drug interactions with Rifapentine or INH
* On medications known to cause hepatoxicity and/or neutropenia

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2026-01-16 (Actual); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Rate of adverse events with 1-m INH/RPT/Vit B6 | 28 days
  Treatment discontinuation due to adverse reaction of study drug determined by investigator

SECONDARY OUTCOMES:
Rate of treatment compliance | 28 days
  Percentage of daily dosage taken within the 28 day course
Rate of treatment completion | 28 days
  Completion of 28 day course within a 5 week period

OTHER OUTCOMES:
Rate of reactivation of active tuberculosis | 2 years
  Rate of culture-confirmed tuberculosis disease after completing study regimen
Trough drug concentration | 28 days
  Isoniazid and Rifapentine serum drug concentration
3-hour post-dose drug concentration | 28 days
  Isoniazid and Rifapentine serum drug concentration

CONTACTS AND LOCATIONS:
Overall Officials: Pinki Bhatt, MD, Principal Investigator — Rutgers
Locations (1):
- Pinki J Bhatt, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Singh N, Paterson DL. Mycobacterium tuberculosis infection in solid-organ transplant recipients: impact and implications for management. Clin Infect Dis. 1998 Nov;27(5):1266-77. doi: 10.1086/514993. PMID 9827281
- [Background] Subramanian A, Dorman S; AST Infectious Diseases Community of Practice. Mycobacterium tuberculosis in solid organ transplant recipients. Am J Transplant. 2009 Dec;9 Suppl 4:S57-62. doi: 10.1111/j.1600-6143.2009.02894.x. No abstract available. PMID 20070696
- [Background] Adamu B, Abdu A, Abba AA, Borodo MM, Tleyjeh IM. Antibiotic prophylaxis for preventing post solid organ transplant tuberculosis. Cochrane Database Syst Rev. 2014 Mar 4;2014(3):CD008597. doi: 10.1002/14651858.CD008597.pub2. PMID 24590589
- [Background] Agarwal SK, Gupta S, Dash SC, Bhowmik D, Tiwari SC. Prospective randomised trial of isoniazid prophylaxis in renal transplant recipient. Int Urol Nephrol. 2004;36(3):425-31. doi: 10.1007/s11255-004-6251-6. PMID 15783119
- [Background] Rafiei N, Williams J, Mulley WR, Trauer JM, Jenkin GA, Rogers BA. Mycobacterium tuberculosis: Active disease and latent infection in a renal transplant cohort. Nephrology (Carlton). 2019 May;24(5):569-574. doi: 10.1111/nep.13386. PMID 29660203
- [Background] van den Boogaard J, Kibiki GS, Kisanga ER, Boeree MJ, Aarnoutse RE. New drugs against tuberculosis: problems, progress, and evaluation of agents in clinical development. Antimicrob Agents Chemother. 2009 Mar;53(3):849-62. doi: 10.1128/AAC.00749-08. Epub 2008 Dec 15. No abstract available. PMID 19075046
- [Background] Zhang T, Zhang M, Rosenthal IM, Grosset JH, Nuermberger EL. Short-course therapy with daily rifapentine in a murine model of latent tuberculosis infection. Am J Respir Crit Care Med. 2009 Dec 1;180(11):1151-7. doi: 10.1164/rccm.200905-0795OC. Epub 2009 Sep 3. PMID 19729664
- [Background] Holland DP, Sanders GD, Hamilton CD, Stout JE. Potential economic viability of two proposed rifapentine-based regimens for treatment of latent tuberculosis infection. PLoS One. 2011;6(7):e22276. doi: 10.1371/journal.pone.0022276. Epub 2011 Jul 18. PMID 21789248
- [Background] Swindells S, Ramchandani R, Gupta A, Benson CA, Leon-Cruz J, Mwelase N, Jean Juste MA, Lama JR, Valencia J, Omoz-Oarhe A, Supparatpinyo K, Masheto G, Mohapi L, da Silva Escada RO, Mawlana S, Banda P, Severe P, Hakim J, Kanyama C, Langat D, Moran L, Andersen J, Fletcher CV, Nuermberger E, Chaisson RE; BRIEF TB/A5279 Study Team. One Month of Rifapentine plus Isoniazid to Prevent HIV-Related Tuberculosis. N Engl J Med. 2019 Mar 14;380(11):1001-1011. doi: 10.1056/NEJMoa1806808. PMID 30865794